CLINICAL TRIAL: NCT02012933
Title: 3,4-Diaminopyridine for Lambert-Eaton Myasthenic Syndrome and Congenital Myasthenia
Brief Title: 3,4-Diaminopyridine for Lambert-Eaton Myasthenic Syndrome (LEMS) and Congenital Myasthenia (CM)
Status: No longer available | Type: Expanded Access
Sponsor: Oregon Health and Science University (Other)
Collaborators: Jacobus Pharmaceutical (Industry)
Responsible Party: Sponsor
Other Study IDs: Jacobus compassionate program
Record Dates: First submitted 2013-12-11; First posted 2013-12-17 (Estimated); Last update posted 2019-12-11 (Actual); Status verified 2019-12

CONDITIONS: Lambert-Eaton Myasthenic Syndrome (LEMS); Congenital Myasthenia (CM)
Keywords: 3,4DAP, LEMS, CM
MeSH Terms: conditions — Lambert-Eaton Myasthenic Syndrome; Myasthenic Syndromes, Congenital | interventions — Amifampridine

INTERVENTIONS:
Drug: 3,4-diaminopyridine — 10mg tablets for up to 100mg per day
  Other Names: 3,4DAP

SUMMARY:
Lambert-Eaton Myasthenic Syndrome (LEMS) is a rare autoimmune disorder which affects the nerve-muscle junction. The major symptoms of LEMS are progressive muscle weakness. Many patients experience other symptoms like dry mouth or impotence. Congenital Myasthenia (CM) is an inherited disorder with similar affects and symptoms.

3,4-Diaminopyridine (DAP) is an experimental drug that has improved strength in some subjects with (LEMS). There are no other accepted treatments for LEMS and DAP has relatively few side effects.

DETAILED DESCRIPTION:
Subjects with clinically confirmed LEMS or CM will receive 3,4-diaminopyridine (3,4 DAP) by mouth in slowly increasing doses. Treatment will begin with 5-10 mg three times a day. A common final dosage is 15-20 mg four or five times a day, as clinically needed, and if tolerated. The upper limit is a total of 100 mg/day. Subjects will be monitored for strength and side effects via routine clinic visits at intervals of one month for the first three months, then every three months for the first year, and at least every six months thereafter. Treatment will be continued indefinitely if a good clinical response is achieved and side effects are tolerable.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of LEMS or CM
* If female and over the age of 9, must have a negative pregnancy test, and, if premenopausal, must be willing to practice an effective form of birth control.
* Must be tested and found by ECG not to have a prolonged Q-Tc syndrome.
* Must agree to have a second ECG at the time of peak drug effect.

Exclusion Criteria:

* Known to have sensitivity to 3,4-DAP
* History of clinical seizures or evidence of seizure activity on screening EEG
* History of severe asthma

Min Age: 2 Years | Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States